CLINICAL TRIAL: NCT03316846
Title: Tailored Internet-delivered Cognitive Behavioral Therapy for Patients With Chronic Pain and Comorbid Psychiatric Distress
Brief Title: Internet-delivered Cognitive Behavioral Therapy for Patients With Chronic Pain and Psychiatric Distress
Acronym: TIPPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140371
Record Dates: First submitted 2017-09-01; First posted 2017-10-20 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Chronic Pain; Depressive Symptoms; Anxiety; Stress, Psychological
Keywords: Chronic Pain; Depression; Anxiety; Stress; iCBT; Cognitive behavioral therapy; Internet delivered; Tailored treatment
MeSH Terms: conditions — Chronic Pain; Depression; Anxiety Disorders; Stress, Psychological

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-delivered therapy (Experimental): 10 week, guided and individually tailored internet-delivered cognitive behavioral therapy.
  Interventions: Behavioral: Internet-Delivered Cognitive Behavioral Therapy
- Wait list control group (No Intervention): Wait list control group, receives treatment at later point.

INTERVENTIONS:
Behavioral: Internet-Delivered Cognitive Behavioral Therapy
  Arms: Internet-delivered therapy

SUMMARY:
This study is a randomized controlled trial studying the efficacy of an iCBT treatment for patients with chronic pain and comorbid psychiatric distress. Half the participants will receive treatment at first, while the other half serve as a control group. After the first group has received treatment, the same program will be offered to participants in the control group. Treatment will be tailored on the level of individual participants, enabling individuals suffering a wide range of problems to be recruited. The treatment will consist of a 10-week guided self-help program, followed by a booster program and follow-up one year later. During the curse of the treatment the participants will be guided via text communication by a licensed psychologist or a candidate psychologist on their last year of studies.

The primary hypothesis is that an individually tailored CBT-treatment administered through the internet can be beneficial for patients suffering from chronic pain and comorbid psychiatric distress. The investigators expect that patients in the treatment group will show reduced levels of disability, depression and anxiety, while improving on scales measuring coping and quality of life.

DETAILED DESCRIPTION:
Patients suffering from chronic pain often experience comorbid psychiatric distress. Cognitive behavioral therapy (CBT) has been shown to be effective in treating both these problems. However delivering relevant treatment can be difficult due to logistics, cost and lack of personnel with required competence. Delivering CBT though the internet (iCBT) is a novel approach, sidestepping logistical issues while lowering costs. This however, is an area were research is lacking, and though there are several studies showing iCBT to be efficacious in treating both pain and psychiatric conditions, research on a combined approach is scarce.

This study will primarily investigate whether an individually tailored CBT-treatment administered through the internet can be beneficial for patients suffering from chronic pain and comorbid psychiatric conditions. The project will also clarify whether a following booster-program, also administered tough the internet, is helpful in maintaining and increasing effects of the initial treatment. Lastly, analysis of possible mediating variables will be able to give insight into the internal workings of the treatment itself, further elucidating efficacy of specific interventions, data which will be useful in future developments of treatment design.

The treatment will be based on a previously developed program, devised to target depression and anxiety in patients with chronic pain. The treatment will consist of a 10-week period where participants would get access to a series of treatment modules, each addressing a separate problem area using CBT techniques. The treatment includes modules addressing depression, anxiety, panic, worry, insomnia, stress, trauma, communication skills, and relaxation. The booster program will be based on the initial treatment, but will shorter, focusing on repetition, strategies for maintenance, and coping with setbacks. The platform used is an existing platform employed by Smärtcentrum at Uppsala university hospital for delivering internet based treatments.

The study will be conducted using a randomized controlled trial with a between-group design. Participants will be randomized to two groups, were one group will gain access to iCBT treatment while the second group will be a wait-list control, and will gain access to the program once treatment of the active group is finished. Participants will assessed by a licensed psychologist, and treatment modules assigned based on their individual needs. In addition to online CBT modules, consisting of information, exercises and homework assignments, all participants will have regular contact by secure email-channel with a licensed psychologist or last-year psychology student under supervision. This contact will guide treatment, providing support, feedback on homework, and if necessary clarify treatment content and help with IT-related problems interfering with treatment adherence. After a year, participants will be invited to take part in a follow-up module, consisting of limited treatment recapitulation and evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Experienced pain for at least the three previous months
* Medically evaluated regarding the pain condition
* Experiences at least one type of psychological distress such as: depression, anxiety, insomnia or stress
* Access to, and ability to use, a personal computer with internet access
* Mastery of the swedish language

Exclusion Criteria:

* Currently undergoing or planning to undergo CBT-treatment during the course of the study
* Currently undergoing or planning to undergo major changes in pharmacotherapy during the course of the study, or have made such changes in the last 2 months
* Have planned surgical intervention during the course of the study
* Currently experiencing symptoms of severe depression (scores >16 on suicidality on M.I.N.I.)
* Currently experiencing significant symptoms of psychosis (fulfills M.I.N.I criteria for psychotic syndrome, current)
* Currently experiencing significant symptoms of alcohol or substance abuse (fulfills M.I.N.I criteria for alcohol- or substance use disorder)

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in depressive symptoms | at 10 weeks
  Self reported change in depressive symptoms, Montgomery-Åsberg Depression Rating Scale (MADRS-S) Swedish version, 9 items
Change from baseline in depressive symptoms | at one-year
  Self reported change in depressive symptoms, Montgomery-Åsberg Depression Rating Scale (MADRS-S) Swedish version, 9 items
Change from baseline in psychosocial consequences of pain | at 10 weeks
  Self reported psychosocial consequences of pain, West Haven-Yale Multidimensional Pain Inventory (WHY/MPI-S part 1), Swedish version, 22 items
Change from baseline in psychosocial consequences of pain | at one-year
  Self reported psychosocial consequences of pain, West Haven-Yale Multidimensional Pain Inventory (WHY/MPI-S part 1), Swedish version, 22 items

SECONDARY OUTCOMES:
Change from baseline in anxiety sensitivity | at 10 weeks
  Self reported anxiety sensitivity, Anxiety Sensitivity Index (ASI), Swedish version, 16 items
Change from baseline in anxiety sensitivity | at one-year
  Self reported anxiety sensitivity, Anxiety Sensitivity Index (ASI), Swedish version, 16 items
Change from baseline in symptoms of depression and anxiety | at 10 weeks
  Self reported symptoms of depression and anxiety, Hospital Anxiety and Depression Scale (HADS), Swedish version, 14 items
Change from baseline in symptoms of depression and anxiety | at one-year
  Self reported symptoms of depression and anxiety, Hospital Anxiety and Depression Scale (HADS), Swedish version, 14 items
Change from baseline in pain disability | at 10 weeks
  Self reported pain disability, Pain Disability Index (PDI), Swedish version, 7 items
Change from baseline in pain disability | at one-year
  Self reported pain disability, Pain Disability Index (PDI), Swedish version, 7 items
Change from baseline in quality of life | at 10 weeks
  Self reported quality of life, Quality of Life Inventory (QOLI), Swedish version, 7 items
Change from baseline in quality of life | at one-year
  Self reported quality of life, Quality of Life Inventory (QOLI), Swedish version, 7 items
Fear of pain due to movement | Baseline only
  Self reported fear of movement, Tampa Scale of Kinesiophobia (TSK), Swedish version, 17 items
Change from baseline in insomnia symptoms | at 10 weeks
  Self reported insomnia symptoms, Insomnia Severity Index (ISI), Swedish version
Change from baseline in insomnia symptoms | at one-year
  Self reported insomnia symptoms, Insomnia Severity Index (ISI), Swedish version
Change from baseline in PTSD symptoms | at 10 weeks
  Self reported PTSD symptoms, Post-Traumatic Stress Disorder checklist 5 (PCL-5), Swedish version
Change from baseline in PTSD symptoms | at one-year
  Self reported PTSD symptoms, Post-Traumatic Stress Disorder checklist 5 (PCL-5), Swedish version
Change from baseline in stress | at 10 weeks
  Self reported stress, Shirom-Melomed Burnout Questionnaire (SMBQ), Swedish version
Change from baseline in stress | at one-year
  Self reported stress, Shirom-Melomed Burnout Questionnaire (SMBQ), Swedish version
Change from baseline in GAD-symptoms | at 10 weeks
  Self reported GAD-symptoms , Generalized Anxiety Disorder 7 (GAD-7), Swedish version
Change from baseline in GAD-symptoms | at one-year
  Self reported GAD-symptoms , Generalized Anxiety Disorder 7 (GAD-7), Swedish version
Change from baseline in pain catastrophizing | at 5 weeks
  Self reported pain catastrophizing, Pain Catastrophizing Scale (PCS), Swedish version
Change from baseline in pain catastrophizing | at 10 weeks
  Self reported pain catastrophizing, Pain Catastrophizing Scale (PCS), Swedish version
Change from baseline in pain catastrophizing | at one-year
  Self reported pain catastrophizing, Pain Catastrophizing Scale (PCS), Swedish version
Change from baseline in coping strategies | at one-year
  Self reported coping strategies , Coping Strategies Questionnaire - Revised (CSQ-R), Swedish version
Change from baseline in coping strategies | at 5 weeks
  Self reported coping strategies , Coping Strategies Questionnaire - Revised (CSQ-R), Swedish version
Change from baseline in coping strategies | at 10 weeks
  Self reported coping strategies , Coping Strategies Questionnaire - Revised (CSQ-R), Swedish version
Change from baseline in pain acceptance | at 5 weeks
  Self reported pain acceptance, Chronic Pain Acceptance Questionnaire (CPAQ), Swedish version
Change from baseline in pain acceptance | at 10 weeks
  Self reported pain acceptance, Chronic Pain Acceptance Questionnaire (CPAQ), Swedish version
Change from baseline in pain acceptance | at one-year
  Self reported pain acceptance, Chronic Pain Acceptance Questionnaire (CPAQ), Swedish version
Change from baseline in self efficacy | at 5 weeks
  Self reported pain related self efficacy, Pain Self Efficacy-2 (PSEQ-2), Swedish version
Change from baseline in self efficacy | at 10 weeks
  Self reported pain related self efficacy, Pain Self Efficacy-2 (PSEQ-2), Swedish version
Change from baseline in self efficacy | at one-year
  Self reported pain related self efficacy, Pain Self Efficacy-2 (PSEQ-2), Swedish version
Treatment credibility rating | Baseline only
  Self reported treatment credibility, Treatment Credibility Scale (TCS), Swedish version

CONTACTS AND LOCATIONS:
Overall Officials: Monica Buhrman, PhD, Study Director — Uppsala University; Gerhard Andersson, Professor, Study Chair — Linkoeping University; Torsten Gordh, Professor, Study Chair — Uppsala University
Locations (1):
- Department of Psychology, Uppsala University, Uppsala, Uppland, Sweden